CLINICAL TRIAL: NCT01713361
Title: An Open-label, Randomized, Active Comparator-Controlled, Adaptive Parallel-group Phase 2 Study to Assess the Safety and Efficacy of Multiple Doses of ISIS 416858 Administered Subcutaneously to Patients Undergoing Total Knee Arthroplasty
Brief Title: Active Comparator-Controlled Study to Assess Safety and Efficacy of ISIS-FXIRx in Total Knee Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ISIS 416858-CS3
Record Dates: First submitted 2012-10-04; First posted 2012-10-24 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Venous Thromboembolism
Keywords: total knee arthroplasty; Prophylaxis
MeSH Terms: conditions — Venous Thromboembolism | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ISIS-FXIRx Dose 2 (Experimental): Group B: ISIS-FXIRx Dose #2
  Interventions: Drug: ISIS-FXIRx Dose #2
- ISIS-FXIRx Dose 3 (Experimental): Group C: ISIS-FXIRx Dose #3
  Interventions: Drug: ISIS-FXIRx Dose #3
- Enoxaparin (Active Comparator): Enoxaparin (40mg)
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: ISIS-FXIRx Dose #2 — Group B: ISIS-FXIRx dose #2 subcutaneously administered 7 times prior to total knee arthroplasty, and 2 times after surgery.
  Other Names: ISIS-FXIRx
  Arms: ISIS-FXIRx Dose 2
Drug: ISIS-FXIRx Dose #3 — Group C: ISIS-FXIRx dose #3 subcutaneously administered 7 times prior to total knee arthroplasty, and 2 times after surgery.
  Other Names: ISIS-FXIRx
  Arms: ISIS-FXIRx Dose 3
Drug: Enoxaparin — Enoxaparin (40mg) will be administered by subcutaneous injection the evening prior to total knee arthroplasty (optionally), 6 to 8 hours after surgery, followed by daily injections for at least 8 additional days post surgery (a total of at least 9 consecutive days). [Except for Canadian region, in which the subcutaneous injection of enoxaparin the evening prior to total knee arthroplasty is expected, resulting in a total of at least 10 consecutive days of enoxaparin.]
  Other Names: Lovenox; Clexane
  Arms: Enoxaparin

SUMMARY:
The purpose of this study is:

* To assess the safety and efficacy profile of ISIS-FXIRx, including incidence of bleeding and VTE, in patients undergoing total knee arthroplasty.
* To compare the efficacy and safety profile of ISIS-FXIRx in patients who achieve less than or equal to 0.2 U/mL FXI activity levels to that of enoxaparin.

ELIGIBILITY:
Inclusion Criteria:

* Give written informed consent
* Females must be non-pregnant and non-lactating, and either surgically sterile or post-menopausal. Males must be surgically sterile, abstinent, or if engaged in sexual relations of child-bearing potential, must use contraception
* Undergoing elective, primary unilateral total knee arthroplasty

Exclusion Criteria:

* Body weight <50 kg
* Patients at increased risk of bleeding. History of intracranial or intraocular bleeding. History of gastrointestinal and/or endoscopically verified ulcer disease within the past year.
* History of excessive intra- or direct post operative bleeding or a traumatic spinal or epidural anesthesia
* Brain, spinal, or ophthalmologic surgery within the past 3 months
* History of clinically significant liver disease in the past year
* Screening laboratory results as follows, or any other clinically significant abnormalities in screening laboratory values

  * aPTT or PT or INR >ULN
  * Factor IX activity <LLN
  * Factor VIII activity, vWF antigen or Ristocetin cofactor activity <0.5 U/mL
  * FXI activity <0.3 U/mL
  * Urine protein or blood persistently positive by dipstick. In the event of positive test results, eligibility may be confirmed with urine microscopy or 24 hour urine protein measurement as applicable
  * ALT or AST >1.5 x ULN
  * Total bilirubin >ULN
  * Platelet count <150,000 (or history of thrombocytopenia)
* Hypersensitivity to enoxaparin
* Anticipated concomitant use of anticoagulants/antiplatelet agents or the NSAID nimesulide that may affect study outcome or any other drug influencing coagulation (except low dose aspirin and short acting NSAIDs with a half-life <20 hours) at least 7 days before surgery or during treatment with ISIS Rx.
* Anticipated use of indwelling intrathecal or epidural catheters
* Anemia at Screening
* Have any other conditions which could interfere with the patient participating in or completing the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Primary efficacy outcome | up to 12 days post-surgery
  Composite of asymptomatic DVT (via bilateral venography), and symptomatic VTE, fatal PE, and unexplained death.

SECONDARY OUTCOMES:
Secondary efficacy outcome | 1st dose to up to Day 76
  All DVTs and PEs up to 4 weeks after bilateral venography

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Bhanot, MD, PhD, Study Director — VP, Clinical Development, Isis Pharmaceuticals
Locations (19):
- Bulgaria (3):
  - Isis Investigational Site, Plovdiv
  - Isis Investigational Site, Rousse
  - Isis Investigational Site, Sofia
- Canada (2):
  - Isis Investigational Site, Ajax, Ontario
  - Isis Investigational Site, Oshawa, Ontario
- Latvia (3):
  - Isis Investigational Site, Ādaži
  - Isis Investigational Site, Riga
  - Isis Investigational Site, Valmiera
- Russia (5):
  - Isis Investigational Site, Chelyabinsk
  - Isis Investigational Site, Orenburg
  - Isis Investigational Site, Saint Petersburg
  - Isis Investigational Site, Samara
  - Isis Investigational Site, Yaroslavl
- Ukraine (6):
  - Isis Investigational Site, Cherkassy
  - Isis Investigational Site, Ivano-Frankivsk
  - Isis Investigational Site, Kharkiv
  - Isis Investigational Site, Kyiv
  - Isis Investigational Site, Odesa
  - Isis Investigational Site, Sevastopol

REFERENCES:
- [Derived] Buller HR, Bethune C, Bhanot S, Gailani D, Monia BP, Raskob GE, Segers A, Verhamme P, Weitz JI; FXI-ASO TKA Investigators. Factor XI antisense oligonucleotide for prevention of venous thrombosis. N Engl J Med. 2015 Jan 15;372(3):232-40. doi: 10.1056/NEJMoa1405760. Epub 2014 Dec 7. PMID 25482425